CLINICAL TRIAL: NCT02907385
Title: Efficacy and Safety of LifeSeal™ Kit for Staple Line Sealing in Colorectal and Coloanal Anastomoses: A Prospective Randomized Study
Brief Title: Efficacy and Safety of LifeSeal™ Kit for Colorectal Staple Line Sealing
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LifeBond Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLP-LS-0131
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Rectal Cancer; Anastomotic Leak
Keywords: Rectal Cancer; Low Anterior Resection; LifeSeal; Surgical Sealant
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LifeSeal™ Kit (Experimental): Stapled Anastomosis is performed according to Standard of Care (SoC) with the addition of LifeSeal™ Kit application during surgery.
  Interventions: Device: LifeSeal™ Kit
- Standard of Care (No Intervention): Stapled Anastomosis is performed according to SoC without LifeSeal™ reinforcement.

INTERVENTIONS:
Device: LifeSeal™ Kit — LifeSeal™ Kit is applied as an additional protective layer over a stapled anastomosis
  Arms: LifeSeal™ Kit

SUMMARY:
LifeSeal™ Kit, surgical sealant designed for staple-line reinforcement that is applied over the anastomotic line to prevent bowel content leakage until full physiological function is restored.

RATIONALE : Postoperative anastomotic leakage is one of the most devastating and feared complications in colorectal surgery. The risk of postoperative anastomotic leakage varies widely depending on the level of anastomosis while the risk is higher in low anastomosis.

In order to best demonstrate the benefits of LifeSeal™ in providing staple line reinforcement and helping to reduce leaks, the study includes high risk anastomoses, defined as colorectal and coloanal anastomoses performed within 10 cm from the anal verge.

STUDY DESIGN: This study is designed as a prospective, multi-center, multinational randomized, single-blind, double armed study PRIMARY OBJECTIVE: The primary objective of this study is to assess the efficacy and safety of LifeSeal™ Kit as measured by the change in overall anastomotic leak rates in subjects undergoing low anterior resection with an anastomosis below 10 cm from the anal verge, over the first 17 weeks after surgery.

SECONDARY OBJECTIVES: The secondary objective of this study is to assess the incidence of post-operative leaks and additional benefits that could be related to the use of LifeSeal™ Kit such as reducing the severity and improving the outcome of a leak once it has occurred. In addition, the study will allow for collection and analysis of additional safety data and usability assessment of the device, medical resource utilization, and health related quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 21 years of age at Screening Visit.
2. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
3. Subject is diagnosed with colorectal cancer
4. Subject is scheduled for elective open, laparoscopic or robot assisted surgery involving the creation of a circular stapled anastomosis created within 10cm from the anal verge.
5. Procedure involving Total Mesorectal Excision by an abdominal or transanal approach.
6. Female subjects in child bearing age must be using acceptable contraception methods such as hormonal contraception or two forms of barrier contraception. Acceptable contraception must be used consistently from 30 days before screening until 3 years following surgery

Exclusion Criteria:

Pre-operative exclusion criteria:

1. Female subject who is pregnant, breastfeeding, or if of child bearing potential is unwilling to practice birth control until 3 years following surgery.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
3. Subject has a history of hypersensitivity to porcine derived gelatin or collagen.
4. Subject has a history of hypersensitivity to microbial Transglutaminase.
5. Subject has a known dysfibrinogenemia, hypofibrinogenemia or a fibrinogenemia, without preoperative correction of fibrinogen levels.
6. Subject participating in any other study involving an investigational (unapproved) drug or device within the past 60 days.
7. Subject participating in studies involving approved drug or device will be enrolled only following a mutual consideration of the investigator together with the Sponsor.
8. Subject with a BMI ≥50, which may interfere with access to the surgical site and increase overall operative risk.
9. Subject with American Society of Anesthesiology (ASA) status higher than 3.
10. Avastin use within 30 days prior to surgery.
11. Subject who has undergone a prior pelvic anastomosis.
12. Subject is scheduled for another surgery during the first 6 months following surgery (not including stoma closure ,placement of port for chemotherapy or ureter stent insertion).
13. Subject with an active abdominal or pelvic infection at the operation site.
14. Subject has been previously treated with LifeSeal™ Surgical Sealant.

Intra-operative Exclusion Criteria

1. Anastomosis or procedure (TME) was performed differently from what was defined in the inclusion criteria.
2. Subject received intra-operative sealant, glue or any buttressing material other than the LifeSeal™ Surgical Sealant.
3. Subject has peritoneal carcinomatosis.
4. Subject requires additional unrelated anastomosis during the surgery.
5. Subject is going through another surgical procedure (other than ileostomy or adhesiolysis) during the surgery.
6. Excessive bleeding (above 500cc) identified prior to anastomosis formation with the need for intra-operative blood transfusion.

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of overall anastomotic leak | Up to 17 weeks post surgery

SECONDARY OUTCOMES:
Incidence of post operative anastomotic leaks | Up to 17 weeks post surgery

CONTACTS AND LOCATIONS:
Locations (39):
- United States (23):
  - University of Southern CA, Los Angeles, California
  - Stanford University, Stanford, California
  - Florida Hospital, Florida City, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - University of Chicago, Chicago, Illinois
  - Franciscan, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, Jefferson, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Medical University SC (MUSC), Worcester, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Albany medical center, Albany, New York
  - New York University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Penn state university, State College, Pennsylvania
  - Duke University, Durham, South Carolina
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (4):
  - OLV Ziekenhuis Aalst, Aalst
  - Ziekenhuis Oost-Limburg, Genk
  - Gent University Hospital, Ghent
  - University Hospital Leuven, Leuven
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Zealand University Hospital, Roskilde
- Israel (3):
  - Beilinson Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (3):
  - Policlinico S.Orsola Malpighi, Bologna
  - Humanitas Research Hospital, Milan
  - University of Padova, Padua
- Catharina Hospital Eindhoven, Eindhoven, Netherlands
- Sweden (3):
  - Lund University Hospital, Malmo
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala